CLINICAL TRIAL: NCT01765803
Title: A Single Institution Feasibility Study to Assess Thioridazine as a Mobilizing Agent for CD34+ Hematopoietic Progenitor Cells
Brief Title: Feasibility of Thioridazine as a Mobilizing Agent for CD34+ Hematopoietic Progenitor Cells
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Primary objective not met after planned interim analysis
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Oxnard Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: INST 1208
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Subjects
Keywords: Mellaril; Thioridazine; CD34+; Stem cells; Progenitor cells; Peripheral blood; mobilization; circulation
MeSH Terms: interventions — Thioridazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mellaril (thioridazine) (Experimental): A single 50 gm dose of thioridizine (Mellaril) will be given orally at the beginning of the study
  Interventions: Drug: Mellaril

INTERVENTIONS:
Drug: Mellaril — Subjects will undergo a physical exam including an electrocardiogram (EKG) and have blood drawn before treatment. A single 50 gm dose of thioridazine (Mellaril) will be given to eligible subjects. A second blood draw will occur at 24 hours post-treatment.
  Other Names: Thioridazine

SUMMARY:
This study will investigate the possibility of using the drug thioridazine (also called Mellaril) to increase the number of certain types of cells moving from the bone marrow to the circulation in a group of healthy humans. The types of cells we hope to collect are called CD34+ progenitor, or stem cells. These cells can be used in the laboratory to better understand a number of diseases and suggest new strategies for therapy. Perhaps the most important potential application of human stem cells is the generation of cells and tissues that could be used for cell-based therapies, as a renewable source of replacement cells and tissues to treat diseases including Alzheimer's diseases, spinal cord injury, stroke, burns, heart disease, diabetes, osteoarthritis, and rheumatoid arthritis.

DETAILED DESCRIPTION:
This is a single-arm, feasibility study to test whether a single dose of Mellaril (thioridazine HCL) is able to effectively mobilize CD34+ cells in a set of health human subjects. This study does not involve the use of placebos, and subjects will serve as their own controls for CD34+ cell mobilization. We hypothesize that a single dose of Mellaril (thioridazine HCL) will mobilize CD34+ progenitor cells into human peripheral blood by a factor of at least 10 fold, from 4 to 40 cells/microliter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking subjects (male or female)
* Age: 18 to 55 years
* All subjects must agree to refrain from consuming alcohol during for 48 hours after taking thioridazine.
* Performance status Karnofsky score of 100%.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having not undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* Has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand the purpose and procedures of this study, and the willingness to sign a written informed consent document.
* Only subjects whose laboratory testing, including platelet counts and transaminase levels are within normal limits are eligible.
* Subjects must pass pre-treatment screening by EKG to rule out long QT syndrome or subclinical cardiac arrhythmia.

Exclusion Criteria:

* Subjects who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Agent(s) or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, a febrile illness within 35 days of study entry, or psychiatric illness or dementia, or social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Concomitant use of phenytoin excludes potential subjects from participation.
* Subjects with known long QT syndrome or known history of cardiac arrhythmias are excluded from participation.
* Subjects taking drugs known to inhibit P450 CYP2D6 are excluded from participation.
* Subjects who received an investigational agent within 28 days of dosing with thioridazine on this protocol are excluded from participation.
* Subjects who received thioridazine within 7 days of dosing on this protocol are excluded from participation.
* Subjects who have had pelvic radiation are excluded from participation.
* Subjects who have received myeloablative regimens at any time are excluded from participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart S Winter, MD, Principal Investigator — University of New Mexico Health Sciences Center/Pediatric Oncology
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org
- See also: UNM Cancer Center — http://www.cancer.unm.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mellaril (Thioridazine)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mellaril (Thioridazine)
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 34 [24 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: CD34+ Progenitor Cell Mobilization
Description: To measure CD34+ cells, a peripheral blood draw is taken from the enrolled subject at hour zero on day one of the study before treatment with oral thioridazine. Following treatment, blood draws are taken at 2, 4, 8 and 24 hours. These blood samples are analyzed using Clinical Laboratory Improvement Amendments (CLIA)-approved flow cytometry for CD34+ cell content. CD34+ cell levels will be reported as a percentage of total white blood cells (WBC) in the blood specimens and the difference between baseline and 8 hours will be reported
Time Frame: 8 hours following treatment
Measure: Mean (Standard Deviation); unit: percentage of total WBC count
Arm/Group | Mellaril (Thioridazine)
Number analyzed (Participants) | 6
percentage of total WBC count
  CD34+ cells at baseline | 0.05 (0.015)
  CD34+ cells at 8 hours | 0.05 (0.018)
  Difference between baseline and 8 hours | 0 (0.011)

2. Secondary Outcome: Toxicity
Description: Toxicity will be evaluated according to the grading system (0-5) NCI CTCAE (Common Terminology Criteria for Adverse Events) version 4.
  Any subject who receives treatment on this protocol will be evaluable for toxicity.
Time Frame: Up to 1 month after treatment
Measure: Number; unit: participants
Arm/Group | Mellaril (Thioridazine)
Number analyzed (Participants) | 6
participants
  Grade 1 somnolence | 4
  Returned to baseline within 24 hours | 4

ADVERSE EVENTS:
Arm/Group | Mellaril (Thioridazine)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mellaril (Thioridazine) (N=6)
Somnolence (Sleepiness) (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes